CLINICAL TRIAL: NCT02261181
Title: Preemptive Treatment With XONRID a Medical Device to Reduce Radiation Induced Dermatitis in Head and Neck Cancer Patients Receiving Curative Treatment
Brief Title: Preemptive Treatment With XONRID to Reduce Radiation Induced Dermatitis in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 52/14
Record Dates: First submitted 2014-09-01; First posted 2014-10-10 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Cancer
Keywords: head neck cancer XONRID radiation induced dermatitis
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XONRID (Experimental): Patients will be treated with XONRID + standard of care (SOC) preemptive treatment adopted during radiation treatment for head and neck cancer patients.
  Patients will be instructed to apply the study cream (XONRID) on the irradiated area two times daily, the first application 1-2 h after the morning radiotherapy session, the second in the evening, starting on the first day of irradiation and continuing until 2 weeks after the completion of the radiation treatments or the development of Grade 3 or 4 skin toxicity. When G3 toxicity will occur the patient will be discontinued from the study medication and the skin toxicity will be managed according to internal guidelines. The use of other topical medications for the treatment of dermatitis will be not permitted during the study.
  Interventions: Device: XONRID

INTERVENTIONS:
Device: XONRID — The patients will be treated with XONRID + standard of care (SOC) preemptive treatment adopted during radiation treatment for head and neck cancer patients. Patients will be instructed to apply the study cream (XONRID) on the irradiated area two times daily, the first application 1-2 h after the morning radiotherapy session, the second in the evening, starting on the first day of irradiation and continuing until 2 weeks after the completion of the radiation treatments or the development of Grade 3 or 4 skin toxicity. When G3 toxicity will occur the patient will be discontinued from the study medication and the skin toxicity will be managed according to internal guidelines.

SUMMARY:
There is a strong need to study products with a preemptive role in radiation dermatitis development, with a trial design taking in account patient subjective evaluation and compliance.

XONRID is a promising device for radiation high grade dermatitis prevention; it is a topical gel that prevents and treats skin symptoms such as erythema, itching, burning sensation and pruritus, induced by radiotherapy or other causes.

DETAILED DESCRIPTION:
The patients will be treated with XONRID + standard of care (SOC) preemptive treatment adopted during radiation treatment for head and neck cancer patients in the Institution.

Patients will be planned to receive Intensity-Modulated Radiotherapy Techniques (IMRT or volumetric modulated radiotherapy, VMAT) with conventional fractionation at total dose of 50-66 GY in postoperative setting and 66-70 Gy in radical setting. Radiotherapy will be planned with simultaneous boost (SIB) approaches, using conventional fractionation (1.8-2.12 Gy/die). According to histology, stage and pathology reports, patients could receive concomitant platinum based chemotherapy.

The patients will be evaluated at baseline, at weekly intervals during RT and six months after treatment completion by 2 different treating physicians for each visit. The evaluation will consist of a physician-assessed toxicity assessment using the Radiation Therapy Oncology Group (RTOG), and patient-reported outcome measured using the Skindex-16 questionnaire.

In addition objective in vivo measurements of skin erythema and pigmentation based on reflectance spectrometry (RS) will be performed.

Measurements will be performed before RT, every 5 RT fractions (once a week) up to the end of RT and 6 months after RT completion (same timing as clinical evaluation). Instrumental RS measurement will be performed at five different fixed regions within the area treated with RT, in any cases only on flat skin regions of the neck in an area corresponding to the second node level and in absence of hair or nevus.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Performance status < 2
* Epithelial carcinoma of oropharynx, nasopharynx, larynx, hypopharynx, paranasal sinus and salivary glands
* Planned to receive at least 50 Gy on one side of the neck with at least the 2nd level of neck nodes irradiated
* Postoperative or curative radiation treatment
* Concurrent platinum based chemotherapy is accepted, but not mandatory
* Conventional fractionation (1.8-2.12 GY per fraction, one daily fraction, 5 fractions a week )

Exclusion Criteria:

* Pregnant or lactating women
* Planned to receive concurrent cetuximab
* Previous radiation therapy on the head and neck area
* Cutaneous and connettive diseases (i.e. lupus erythematosus or scleroderma)
* Systemic diseases known to delay the skin healing process such as diabetes mellitus or severe renal failure.
* Use of a tissue-equivalent bolus
* Use of over-the-counter topical medications containing steroids
* Presence of rashes or unhealed wounds in the radiation field
* Recent sun exposure
* Mental conditions that could adversely affect patients' adherence to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Worst skin toxicity | 14 months
  Worst skin toxicity during treatment and until 2 weeks after according to CTCAE , as assessed independently by 2 physicians

SECONDARY OUTCOMES:
MeanPatient Reported Outcome (PRO) | 14 months
  Mean and worst score (measured on a numeric 0-6 scale, where 0= absence of symptom and 6= worst intensity of symptom) of Patient Reported Outcome (PRO) with Skindex 16 questionnaire performed weekly until reaching a total dose of 50 Gy on neck
Median time to G2 radiation dermatitis development | 14 months
  Median time to G2 radiation dermatitis development according to CTCAE
Compliance | 14 months
  Compliance to experimental treatment assumption considering a complete cpmpliance from 0 to 2 applications skipped, a partial compiance from 3 to 10 applications skipped and an absent compliance from 11 to 14 applications skipped.
Grade of late toxicity | 14 months
  Grade of late toxicity (skin fibrosis according to CTCAE) at 6 month follow up visit after treatment ending

CONTACTS AND LOCATIONS:
Overall Officials: Ester Orlandi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

REFERENCES:
- [Derived] Ingargiola R, De Santis MC, Iacovelli NA, Facchinetti N, Cavallo A, Ivaldi E, Dispinzieri M, Franceschini M, Giandini C, Romanello DA, Di Biaso S, Sabetti M, Locati L, Alfieri S, Bossi P, Guglielmo M, Macchi F, Lozza L, Valdagni R, Fallai C, Pignoli E, Orlandi E. A monocentric, open-label randomized standard-of-care controlled study of XONRID(R), a medical device for the prevention and treatment of radiation-induced dermatitis in breast and head and neck cancer patients. Radiat Oncol. 2020 Aug 13;15(1):193. doi: 10.1186/s13014-020-01633-0. PMID 32791985